CLINICAL TRIAL: NCT00141141
Title: A Phase IV, Multicenter, Randomized, Open Label Study To Evaluate The Efficacy And Safety Of Atorvastatin Versus Simvastatin In Type 2 Diabetic Subjects With Hypercholesterolemia
Brief Title: Efficacy And Safety Study Of Atorvastatin Versus Simvastatin In Type 2 Diabetic Subjects With Hypercholesterolemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2581053
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Atorvastatin; Simvastatin

INTERVENTIONS:
Drug: Atorvastatin
Drug: Simvastatin

SUMMARY:
The purpose of this study is to evaluate the efficacy of Atorvastin vs Simvastatin in decreasing LDL-C in diabetic subjects with hypercholesterolemia at the end of the treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus
* LDL-C > 130 mg/dL

Exclusion Criteria:

* Insulin therapy
* Clinically relevant organ disease (creatininemia >2mg/dL, CHF NYHA III and IV)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2004-01; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the decrease of LDL-C after 24 weeks of treatment.

SECONDARY OUTCOMES:
To evaluate the changes from baseline of targeted blood markers.
To evaluate safety of Atorvastatin vs Simvastatin

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (28):
- Italy (28):
  - Pfizer Investigational Site, S. Benedetto DEL Tronto, Ascoli Piceno
  - Pfizer Investigational Site, S.Pietro Vernotico, Brindisi
  - Pfizer Investigational Site, Casarano, Lecce
  - Pfizer Investigational Site, Pavia, PV
  - Pfizer Investigational Site, Orbassano, Torino
  - Pfizer Investigational Site, Mestre, VE
  - Pfizer Investigational Site, Ancona
  - Pfizer Investigational Site, Asti
  - Pfizer Investigational Site, Bari
  - Pfizer Investigational Site, Cagliari
  - Pfizer Investigational Site, Campobasso
  - Pfizer Investigational Site, Catania
  - Pfizer Investigational Site, Catanzaro
  - Pfizer Investigational Site, Ferrara
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Messina
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Palermo
  - Pfizer Investigational Site, Parma
  - Pfizer Investigational Site, Perugia
  - Pfizer Investigational Site, Pisa
  - Pfizer Investigational Site, Potenza
  - Pfizer Investigational Site, Rimini
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, S. Benedetto Del Tronto (AP)
  - Pfizer Investigational Site, Torino
  - Pfizer Investigational Site, Udine

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581053&StudyName=Efficacy%20And%20Safety%20Study%20Of%20Atorvastatin%20Versus%20Simvastatin%20In%20Type%202%20Diabetic%20Subjects%20With%20Hypercholesterolemia